CLINICAL TRIAL: NCT03539263
Title: Randomized Controlled Experimental Trial Designed to Test the Effects of Probiotics on Mood
Brief Title: Effects of Probiotics on Mood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probiotical S.p.A. (Industry)
Collaborators: Universita di Verona (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 766CESC
Record Dates: First submitted 2018-04-06; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The trial design is parallel, with two groups (experimental group and control group) and four evaluation sessions at intervals of three weeks (T0wk = baseline, T3wk = intermediate, T6wk=final and T9wk = follow-up).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): the subjects are treated with probiotics: Bifihappy
  Interventions: Dietary Supplement: Bifihappy
- Group 2 (Placebo Comparator): the subjects are treated with a placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifihappy — During the six weeks of treatment, the experimental group will take daily doses of 2,5 g with a concentration of 4x109 CFU/sachet of a mixture of lyophilised probiotic strains of the following species:
  * Lactobacillus fermentum
  * Lactobacillus rhamnosus
  * Lactobacillus plantarum
  * Bifidobacterium longum
  Arms: Group 1
Other: Placebo — During the six weeks of treatment, the experimental group will take daily doses of 2,5 g of maltodextrin
  Arms: Group 2

SUMMARY:
Recent demonstration that probiotics administration has positive effects on depressive feelings in healthy populations suggests its possible role as an adjuvant therapy for depression in clinical populations and as a non-invasive strategy to prevent depressive feelings in healthy individuals. The present study extends current knowledge on the beneficial effects of probiotics on psychological well-being, as measured by changes in mood (e.g., depression, anxiety, cognitive reactivity to sad mood), personality dimensions, and quality of sleep, which have been considered as related to mood. For this double-blind, placebo-controlled study healthy volunteers pseudo-randomly assigned to an experimental or control group assumed a daily dose of probiotic or placebo, respectively, for 6 weeks. Mood, personality dimensions, and sleep quality were assessed four times (before the beginning of the study, at 3 and 6 weeks, and at 3 weeks of washout).

DETAILED DESCRIPTION:
A. THEORETICAL BACKGROUND The intestine and the brain are intimately connected with each other through the gut-brain axis, which involves bidirectional communication between the nervous, endocrine and immune systems. In the last years, it has become increasingly evident that this communication implies also interactions with the intestinal bacterial flora, which releases immune activation and other signalling molecules that may play a major role in the regulation of the brain and human behaviour. For instance, the microbiota produces neuroactive substances and their precursors (e.g. tryptophan) that may reach the brain through the endocrine and autonomous nervous system. Recently, the interest has been focused also on the cognitive field. Indeed, there is experimental evidence that bacterial products may positively influence cognitive functions, such as spatial memory and problem-solving abilities. Moreover, probiotics seem to exercise influence on mood, anxiety and depression, opening new therapeutic prospects. A recent trial showed that four weeks of taking probiotics (Bifidobacterium bifidum W23, Bifidobacterium lactis W52, Lactobacillus acidophilus W37, Lactobacillus brevis W63, Lactobacillus casei W56, Lactobacillus salivarius W24, Lactococcus lactis W19 e W58) led to an improvement in mood, fostering reduction in negative thoughts.

B. THE PURPOSE OF THE RESEARCH PROJECT The primary goal of the trial is to investigate the effect of probiotics on depression. Moreover, it will assess also effects on anxiety and other personality traits in healthy young students. The trial intends also to investigate whether probiotics may influence the quality of sleep and bowel habits. The trial will be placebo-controlled, randomized, pre- and post-intervention, double-blind designed (investigator and participants). In the light of the several end-points examined, the statistical analysis will be of explorative type.

The collection of faecal samples will allow, in case of finding any effects of the administered product on mood, to go back to any microbial components that have changed in individuals following the treatment. Monitoring (see below) the normal feed and physical habits of the individuals will allow to check the possible effect of these confounding factors on the parameters measured in the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and Famale subjects.
* Aged between 18 and 35.
* Already owing a smartphone with Android or iOS system.

Exclusion Criteria:

* Drug taking, smoking, coeliac disease, lactose intolerance.
* Disorders such as IBS (Irritable Bowel Syndrome), IBD (Irritable Bowel Disease), UC (Ulcerative Colitis) and other serious diseases, e.g. MS (Multiple Sclerosis) and diabetes (type 1/type 2).
* Oral intake of antibiotics and other medicines on a continuative basis.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-06-15 (Actual); Study Completion 2017-06-15 (Actual)

PRIMARY OUTCOMES:
Change in the psychological profile | four evaluation sessions at intervals of three weeks of probiotic intervention
  The primary outcome is the difference in the scores at the Leiden Index of Depression Sensitivity-Revised test (LEIDS-R) standardized questionnaire between the experimental and control groups. The Leiden Index of Depression Sensitivity-Revised test, LEIDS-R, is a self-report questionnaire that tests cognitive reactivity to sad mood, which is an index of cognitive vulnerability to depression.

SECONDARY OUTCOMES:
Evaluation of mood - State Trait Anxiety Inventory (STAI) standardized questionnarie. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups. The State Trait Anxiety Inventory, STAI, is a self-report questionnaire that measures the presence and severity of current symptoms of anxiety and the propensity to be anxious.
Evaluation of mood - Beck Depression Inventory (BDI-2) standardized questionnarie. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups. The Beck Depression Inventory, BDI-2, is a self-report questionnaire that measures the occurrence and severity of current depressive symptoms.
Evaluation of mood - Profile od Mood State (POMS) standardized questionnarie. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups. The Profile of Mood State, POMS, is a self-report questionnaire that assesses mood.
Evaluation of the quality of sleep. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups in the standardized questionnaire Pittsburgh Sleep Quality Index (PSQI). The Pittsburgh Sleep Quality Index, PSQI, is a self-report questionnaire that assesses sleep quality for the majority of days and nights in the past months.
Evaluation of personality - Temperament and Character Inventory (TCI) standardized questionnarie. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups. The Temperament and Character Inventory, TCI, is a self-report, true-false questionnaire that measures two components of personality: temperament and character.
Evaluation of personality - Cope Orientation to Problem Experienced-New Italian Version (COPE-NIV) standardized questionnarie. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups. The Cope Orientation to Problem Experienced - New Italian Version, COPE-NIV, is a self-report questionnaire that measures coping strategies: the cognitive and behavioral strategies people use to manage stressful situations.
Evaluation of personality - Behavioral Inhibition System and Behavioral Activation System Scale (BIS/BAS) standardized questionnarie. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups. The Behavioral Inhibition and Behavioral Activation Scale, BIS/BAS, is a self-report questionnaire that measures an individual's sensitivity to behavioral inhibition and behavioral activation systems.
Evaluation of personality - Life Orientation Test-revisited (LOT-R) standardized questionnarie. | four evaluation sessions at intervals of three weeks of probiotic intervention
  difference in the scores between the experimental and control groups. The Life Orientation Test-revisited, LOT-R, is a self-report measure of dispositional optimism and pessimism.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Verona, Verona, Italy

IPD SHARING:
Plan to Share IPD: Yes
Study Protocol
Supporting Information: Study Protocol
Time Frame: from April 2018
Access Criteria: Plos One

REFERENCES:
- [Background] Barrett E, Ross RP, O'Toole PW, Fitzgerald GF, Stanton C. gamma-Aminobutyric acid production by culturable bacteria from the human intestine. J Appl Microbiol. 2012 Aug;113(2):411-7. doi: 10.1111/j.1365-2672.2012.05344.x. Epub 2012 Jun 15. PMID 22612585
- [Background] Beck A, Steer R, Brown G (1996). Manual for Beck Depression Inventory II (BDI-II). San Antonio, TX: Psychology Corporation
- [Background] Block J, Kremen AM. IQ and ego-resiliency: conceptual and empirical connections and separateness. J Pers Soc Psychol. 1996 Feb;70(2):349-61. doi: 10.1037//0022-3514.70.2.349. PMID 8636887
- [Background] Bravo JA, Forsythe P, Chew MV, Escaravage E, Savignac HM, Dinan TG, Bienenstock J, Cryan JF. Ingestion of Lactobacillus strain regulates emotional behavior and central GABA receptor expression in a mouse via the vagus nerve. Proc Natl Acad Sci U S A. 2011 Sep 20;108(38):16050-5. doi: 10.1073/pnas.1102999108. Epub 2011 Aug 29. PMID 21876150
- [Background] Bravo JA, Julio-Pieper M, Forsythe P, Kunze W, Dinan TG, Bienenstock J, Cryan JF. Communication between gastrointestinal bacteria and the nervous system. Curr Opin Pharmacol. 2012 Dec;12(6):667-72. doi: 10.1016/j.coph.2012.09.010. Epub 2012 Oct 4. PMID 23041079
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Cloninger CR, Przybeck TR, Svrakic DM, Wetzel RD (1994). The Temperament and Character Inventory (TCI): A Guide to Its Development and Use (St. Louis, MO: Center for Psychobiology of Personality, Washington University).
- [Background] Cryan JF, Dinan TG. Mind-altering microorganisms: the impact of the gut microbiota on brain and behaviour. Nat Rev Neurosci. 2012 Oct;13(10):701-12. doi: 10.1038/nrn3346. Epub 2012 Sep 12. PMID 22968153
- [Background] Curcio G, Tempesta D, Scarlata S, Marzano C, Moroni F, Rossini PM, Ferrara M, De Gennaro L. Validity of the Italian version of the Pittsburgh Sleep Quality Index (PSQI). Neurol Sci. 2013 Apr;34(4):511-9. doi: 10.1007/s10072-012-1085-y. Epub 2012 Apr 13. PMID 22526760
- [Background] Davis MH (1980). A multidimensional approach to individual differences in empathy. JSAS Catalog of Selected Documents in Psychology, 10, 85
- [Background] Desbonnet L, Garrett L, Clarke G, Bienenstock J, Dinan TG. The probiotic Bifidobacteria infantis: An assessment of potential antidepressant properties in the rat. J Psychiatr Res. 2008 Dec;43(2):164-74. doi: 10.1016/j.jpsychires.2008.03.009. Epub 2008 May 5. PMID 18456279
- [Background] Desbonnet L, Garrett L, Clarke G, Kiely B, Cryan JF, Dinan TG. Effects of the probiotic Bifidobacterium infantis in the maternal separation model of depression. Neuroscience. 2010 Nov 10;170(4):1179-88. doi: 10.1016/j.neuroscience.2010.08.005. Epub 2010 Aug 6. PMID 20696216
- [Background] Farma T & Cortinovis I (2001). Un questionario sul "Locus of Control": suo utilizzo nel contesto italiano. Ricerca in Psicoterapia, 1
- [Background] Foster JA, McVey Neufeld KA. Gut-brain axis: how the microbiome influences anxiety and depression. Trends Neurosci. 2013 May;36(5):305-12. doi: 10.1016/j.tins.2013.01.005. Epub 2013 Feb 4. PMID 23384445
- [Background] Fraher MH, O'Toole PW, Quigley EM. Techniques used to characterize the gut microbiota: a guide for the clinician. Nat Rev Gastroenterol Hepatol. 2012 Mar 27;9(6):312-22. doi: 10.1038/nrgastro.2012.44. PMID 22450307
- [Background] GIRVIN GT, STEVENSON JW. Cell free choline acetylase from Lactobacillus plantarum. Can J Biochem Physiol. 1954 Mar;32(2):131-46. No abstract available. PMID 13141176
- [Background] Grenham S, Clarke G, Cryan JF, Dinan TG. Brain-gut-microbe communication in health and disease. Front Physiol. 2011 Dec 7;2:94. doi: 10.3389/fphys.2011.00094. eCollection 2011. PMID 22162969
- [Background] Grossman MI. Neural and hormonal regulation of gastrointestinal function: an overview. Annu Rev Physiol. 1979;41:27-33. doi: 10.1146/annurev.ph.41.030179.000331. No abstract available. PMID 35089
- [Background] Komatsuzaki N, Nakamura T, Kimura T, Shima J. Characterization of glutamate decarboxylase from a high gamma-aminobutyric acid (GABA)-producer, Lactobacillus paracasei. Biosci Biotechnol Biochem. 2008 Feb;72(2):278-85. doi: 10.1271/bbb.70163. Epub 2008 Feb 7. PMID 18256502
- [Background] Kotov RI, Belmman SB, Watson DB (2004). Multidimensional Iowa Suggestibility Scale (MISS) Brief Manual. Stony Brook School of Medicine.
- [Background] Leone L, Pierro A e Mannetti L. (2002). Validità della versione italiana delle scale BIS/BAS di Carver e White (1994): Generalizzabilità della struttura e relazioni con costrutti affini. Giornale Italiano di Psicologia, 2: 413-434.
- [Background] Li W, Dowd SE, Scurlock B, Acosta-Martinez V, Lyte M. Memory and learning behavior in mice is temporally associated with diet-induced alterations in gut bacteria. Physiol Behav. 2009 Mar 23;96(4-5):557-67. doi: 10.1016/j.physbeh.2008.12.004. Epub 2008 Dec 24. PMID 19135464
- [Background] Lombardo C (2008). Adattamento italiano della Multidimensional Perfectionism Scale (MPS). Psicoterapia cognitiva e comportamentale, 14(1):31-46
- [Background] Martinez RC, Cardarelli HR, Borst W, Albrecht S, Schols H, Gutierrez OP, Maathuis AJ, de Melo Franco BD, De Martinis EC, Zoetendal EG, Venema K, Saad SM, Smidt H. Effect of galactooligosaccharides and Bifidobacterium animalis Bb-12 on growth of Lactobacillus amylovorus DSM 16698, microbial community structure, and metabolite production in an in vitro colonic model set up with human or pig microbiota. FEMS Microbiol Ecol. 2013 Apr;84(1):110-23. doi: 10.1111/1574-6941.12041. Epub 2012 Dec 17. PMID 23167835
- [Background] Mayer EA. Gut feelings: the emerging biology of gut-brain communication. Nat Rev Neurosci. 2011 Jul 13;12(8):453-66. doi: 10.1038/nrn3071. PMID 21750565
- [Background] Mayer EA, Knight R, Mazmanian SK, Cryan JF, Tillisch K. Gut microbes and the brain: paradigm shift in neuroscience. J Neurosci. 2014 Nov 12;34(46):15490-6. doi: 10.1523/JNEUROSCI.3299-14.2014. PMID 25392516
- [Background] McNair DM, Lorr M, Droppleman LF (1964). Poms. Profile of Mood States. San Diego: Educational and Industrial Testing Service; ad. it. Firenze: Giunti O.S. Organizzazioni Speciali, 1991.
- [Background] Mitsou EK, Kirtzalidou E, Oikonomou I, Liosis G, Kyriacou A. Fecal microflora of Greek healthy neonates. Anaerobe. 2008 Apr;14(2):94-101. doi: 10.1016/j.anaerobe.2007.11.002. Epub 2007 Dec 3. PMID 18207437
- [Background] Muyzer G, de Waal EC, Uitterlinden AG. Profiling of complex microbial populations by denaturing gradient gel electrophoresis analysis of polymerase chain reaction-amplified genes coding for 16S rRNA. Appl Environ Microbiol. 1993 Mar;59(3):695-700. doi: 10.1128/aem.59.3.695-700.1993. PMID 7683183
- [Background] Özogul F (2004). Production of biogenic amines by Morganella morganii, Klebsiella pneumoniae andHafnia alvei using a rapid HPLC method. Eur Food Res Technol. 219:465-469.
- [Background] Özogul F, Kuley E, Özogul Y, Özogul I (2012). The function of lactic acid bacteria on bio-genic amines production by food-borne pathogens in arginine decarboxylasebroth. Food Sci Technol Res 18:795- 804
- [Background] Pellegrini N, Salvatore S, Valtuena S, Bedogni G, Porrini M, Pala V, Del Rio D, Sieri S, Miglio C, Krogh V, Zavaroni I, Brighenti F. Development and validation of a food frequency questionnaire for the assessment of dietary total antioxidant capacity. J Nutr. 2007 Jan;137(1):93-8. doi: 10.1093/jn/137.1.93. PMID 17182807
- [Background] Pisani P, Faggiano F, Krogh V, Palli D, Vineis P, Berrino F. Relative validity and reproducibility of a food frequency dietary questionnaire for use in the Italian EPIC centres. Int J Epidemiol. 1997;26 Suppl 1:S152-60. doi: 10.1093/ije/26.suppl_1.s152. PMID 9126543
- [Background] Rowatt, E (1948). The relation of pantothcnic acid to acetylcholine formation by a strain of Lactobacillus plantarum. J. Gen. Microbiol. 2. 1, 25-30
- [Background] Saha DC, Reimer RA. Long-term intake of a high prebiotic fiber diet but not high protein reduces metabolic risk after a high fat challenge and uniquely alters gut microbiota and hepatic gene expression. Nutr Res. 2014 Sep;34(9):789-96. doi: 10.1016/j.nutres.2014.08.004. Epub 2014 Aug 23. PMID 25217504
- [Background] Scheier MF, Carver CS, Bridges MW. Distinguishing optimism from neuroticism (and trait anxiety, self-mastery, and self-esteem): a reevaluation of the Life Orientation Test. J Pers Soc Psychol. 1994 Dec;67(6):1063-78. doi: 10.1037//0022-3514.67.6.1063. PMID 7815302
- [Background] Shishov VA, Kirovskaia TA, Kudrin VS, Oleskin AV. [Amine neuromediators, their precursors, and oxidation products in the culture of Escherichia coli K-12]. Prikl Biokhim Mikrobiol. 2009 Sep-Oct;45(5):550-4. Russian. PMID 19845286
- [Background] Sica C., Magni C., Ghisi M., Altoè G., Sighinolfi C., CHiri L.R., Franceschini S. (2008). Cope Orientation to Problems Experienced - Nuova Versione Italiana (COPE-NVI): uno strumento per la misura degli stili di coping. Psicoterapia cognitiva e comportamentale,14 (1):27-53
- [Background] Snart J, Bibiloni R, Grayson T, Lay C, Zhang H, Allison GE, Laverdiere JK, Temelli F, Vasanthan T, Bell R, Tannock GW. Supplementation of the diet with high-viscosity beta-glucan results in enrichment for lactobacilli in the rat cecum. Appl Environ Microbiol. 2006 Mar;72(3):1925-31. doi: 10.1128/AEM.72.3.1925-1931.2006. PMID 16517639
- [Background] Spielberger CD, Gorsuch RL, Lushene R, Vagg PR, Jacobs GA(1983). Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press
- [Background] Steenbergen L, Sellaro R, van Hemert S, Bosch JA, Colzato LS. A randomized controlled trial to test the effect of multispecies probiotics on cognitive reactivity to sad mood. Brain Behav Immun. 2015 Aug;48:258-64. doi: 10.1016/j.bbi.2015.04.003. Epub 2015 Apr 7. PMID 25862297
- [Background] Tsavkelova EA, Botvinko IV, Kudrin VS, Oleskin AV. Detection of neurotransmitter amines in microorganisms with the use of high-performance liquid chromatography. Dokl Biochem. 2000 May-Jun;372(1-6):115-7. No abstract available. PMID 10935181
- [Background] van der Does W, Williams JMG (2003). Leiden Index of Depression Sensitivity - Revised (LEIDS-R). Leiden University.
- [Background] Walker AW, Ince J, Duncan SH, Webster LM, Holtrop G, Ze X, Brown D, Stares MD, Scott P, Bergerat A, Louis P, McIntosh F, Johnstone AM, Lobley GE, Parkhill J, Flint HJ. Dominant and diet-responsive groups of bacteria within the human colonic microbiota. ISME J. 2011 Feb;5(2):220-30. doi: 10.1038/ismej.2010.118. Epub 2010 Aug 5. PMID 20686513
- [Background] Yang J, Fox M, Cong Y, Chu H, Zheng X, Long Y, Fried M, Dai N. Lactose intolerance in irritable bowel syndrome patients with diarrhoea: the roles of anxiety, activation of the innate mucosal immune system and visceral sensitivity. Aliment Pharmacol Ther. 2014 Feb;39(3):302-11. doi: 10.1111/apt.12582. Epub 2013 Dec 5. PMID 24308871